CLINICAL TRIAL: NCT01924182
Title: Post-market Study Evaluating a Treatment Conversion to Low Dose Intrathecal Morphine From Conventional Medical Management for Maintenance of Pain Control and Improvement of Opioid-related Side Effects. (CONVERT Targeted Drug Delivery [TDD])
Brief Title: Intrathecal Morphine Compared to Conventional Medical Management for Pain Control and Opioid-related Side Effects
Acronym: CONVERT-TDD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Amendment changes were significant enough to warrant a new study.
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1664 - CONVERT-TDD
Record Dates: First submitted 2013-08-13; First posted 2013-08-16 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-02

CONDITIONS: Chronic Pain
Keywords: chronic pain; inadequate pain relief; intolerable side effects
MeSH Terms: conditions — Chronic Pain | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IT group (Intrathecal Morphine Sulfate) (Other): SynchroMed Infusion System and Intrathecal Morphine Sulfate
  Interventions: Device: SynchroMed Infusion System and Intrathecal Morphine Sulfate
- Conventional Medical Management (Other): Conventional Medicine, and then SynchroMed Infusion System and Intrathecal Morphine Sulfate
  Interventions: Device: SynchroMed Infusion System and Intrathecal Morphine Sulfate; Other: Conventional Medicine

INTERVENTIONS:
Device: SynchroMed Infusion System and Intrathecal Morphine Sulfate — Following a successful test of Intrathecal Morphine Sulfate, subjects will undergo surgery to implant the drug pump (SynchroMed Infusion System) and spinal catheter. The pump will deliver morphine directly to the spinal cord for pain control.
  Other Names: SynchroMed infusion system; Intrathecal morphine sulfate; Infumorph; Targeted drug delivery; Spinal morphine; Intrathecal morphine
Other: Conventional Medicine — Subjects will continue to use pain medications as prescribed by their doctor.
  Other Names: Standard of Care
  Arms: Conventional Medical Management

SUMMARY:
This study compares two different ways to treat pain. The two ways are:

1. continuing to take current pain medication(s) or
2. receiving morphine, a pain medication from a drug pump (a system to deliver drug to your body) that is implanted.

None of the procedures or products used in this study are experimental. The length the study will be about 25 weeks (between 5½ to 6½ months). The purpose of this study is to compare pain and opioid side effects between people who get a drug pump and people who do not get a drug pump that will stay on their current pain medication treatment.

DETAILED DESCRIPTION:
This was a randomized, controlled, open-label, multi-center, prospective post-market study to assess pain control and opioid-related side effects following a route of delivery change to low dose IT morphine therapy from systemic opioid therapy. Subjects with nonmalignant, chronic, intractable pain who were experiencing inadequate pain relief and/or intolerable side effects from systemic opioid therapy receiving ≤300 mg/day morphine equivalent dose were eligible for screening. Additionally, the subjects had no known history of sleep apnea and were candidates for IT morphine administration via the SynchroMed Infusion System. Subjects must not have previously undergone an intrathecal/epidural trial for pump infusion therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated Medtronic/IRB approved Informed Consent Form and HIPAA Authorization prior to any study procedures being performed
* Willing and able to attend visits and comply with the study protocol
* Willing and able to abstain from alcohol consumption for the study duration
* At least 18 years of age
* Male or non-pregnant, non-lactating female
* Currently receiving </= 300 mg/day morphine equivalent of systemic opioids at screening
* Used a stable dose of opioids (no change in type or prescribed frequency or dose) for 30 days prior to the Screening as documented in the medical history
* Used chronic systemic opioids for at least 6 months prior to Screening as documented in medical history

Per investigator's medical assessment and the subject's medical history, the subject is/has:

* A new candidate for chronic intrathecal drug therapy (including no prior intrathecal/epidural trial for pump infusion therapy)
* A diagnosis of nonmalignant, chronic intractable pain as documented in the medical history
* Medically stable and able to undergo surgery for implantation of the SynchroMed Infusion System
* Completed a psychological evaluation within 6 months prior to Screening

Exclusion Criteria:

* Psychological or other health conditions, financial, and/or legal concerns (within 3 months prior to Screening) that would interfere with the subject's ability to fulfill the requirements of the protocol as per the investigator's opinion
* A history of alcohol abuse or any illicit drug use within 2 years prior to Screening
* A positive urine test for illicit drugs at Screening (Exception: If subject has a physician's prescription for an illicit drug; for example, medical marijuana)
* Known diagnosis of moderate to severe sleep apnea.
* Prescribed Continuous Positive Airway Pressure (CPAP), Adaptive Servo-Ventilation (ASV) therapy or an oral appliance prescribed for the treatment of moderate to severe sleep apnea (current or previous history)
* An active malignancy or has been diagnosed with cancer and has not been in remission for at least 1 year prior to screening
* An implanted electrical stimulation device(s) or if the subject is expected to require one of these during the course of the study
* Planned to enroll or is currently enrolled in another investigational drug or investigational medical device study or has participated in an investigational drug or medical device study within 30 days prior to Screening

Prior to Randomization, a subject will be excluded if:

* Diary does not meet compliance
* Mean diary-reported 12-hour NPRS < 6 (on 0 to 10 scale, as reported over 5 days)
* Positive urine test for alcohol at Baseline
* Negative urine test for opioids at Baseline
* Baseline sleep study (PSG) with SaO2 <=80% for >= 5 consecutive minutes, and/or an Apnea-Hypopnea Index (AHI) >=15.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CONVERT TDD Clinical Research Study Team, Study Director — MedtronicNeuro
Locations (6):
- United States (6):
  - Pain Management Services PC, Homewood, Alabama
  - Napa Pain Institute and Neurovations, Napa, California
  - IPM Medical Group (Interventional Pain Medical Group), Walnut Creek, California
  - Compass Research, Orlando, Florida
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - University of Virginia Pain Management Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seven participants were enrolled (consented).
Pre-assignment Details: Of the 7 participants that were enrolled, 3 met the randomization eligibility and were randomized to the IT Group. Of the 3 participants randomized, 2 were implanted.
Groups:
- IT Group (SynchroMed/Intrathecal Morphine Sulfate): Subjects randomized to the IT group (Intrathecal morphine sulfate/SynchroMed Infusion System) will have a test injection or infusion of intrathecal morphine to check for pain control and make sure there are no negative reactions. If the test is successful, subjects in the IT group will have a pump and spinal catheter implanted. These subjects will stop using all other pain medications and start using only intrathecal morphine for pain control.
  SynchroMed Infusion System and Intrathecal Morphine Sulfate: Following a successful intrathecal test of morphine, IT morphine subjects will undergo surgery to implant the drug pump (SynchroMed) and spinal catheter. The pump will deliver morphine directly to the spinal cord for pain control.
- Conventional Medical Management: Subjects randomized to the CMM group will continue to use pain medications as prescribed by their doctor. Subjects randomized to CMM will be offered the option of pump implant following completion of the 3-month visit.
Period: Overall Study
Arm/Group | IT Group (SynchroMed/Intrathecal Morphine Sulfate) | Conventional Medical Management
Started | 3 | 0
Completed | 2 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IT Group (SynchroMed/Intrathecal Morphine Sulfate) | Conventional Medical Management | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (11.8) |  | 56.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 1 |  | 1
Baseline patient-reported pain diary score [Mean (Standard Deviation); unit: units on a scale] — Average of 5 days of a patient-reported pain diary. The scale ranges from 0 (no pain) to 10 (pain as bad as you can imagine).
  units on a scale | 7.0 (1.4) |  | 7.0 (1.4)
Baseline 23-item toxicity score [Mean (Standard Deviation); unit: units on a scale] — A subset of 23 specific items related to opioid side effects from the Common Terminology Criteria for Adverse Events from the National Cancer Institute. The item scores were summed. The range of the total score is 0 (best case) to 90 (worst case).
  units on a scale | 8.7 (3.8) |  | 8.7 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success
Description: Determine the proportion of subjects with clinical success based on changes in pain intensity (Numerical Pain Rating Scale: NPRS) and opioid-related Common Toxicity Criteria for Adverse Events (CTCAE) from the National Cancer Institute (NCI).
Time Frame: 3 Month
Population: 2 of the 3 randomized participants did not complete the follow-up or provide outcome information. As there was only 1 participant that completed the primary outcome assessment, no statistical analysis will be presented.
Measure: Number; unit: participants
Arm/Group | IT Group (SynchroMed/Intrathecal Morphine Sulfate) | Conventional Medical Management
Number analyzed (Participants) | 1 | 0
participants | 1 |

2. Secondary Outcome: Pain Assessment
Description: Compare changes from Baseline to Month 3 between the IT group and CMM group in Numeric Pain Rating Scale (NPRS). The scale measures pain intensity. Using NPRS, a pain score ranging from 0 (no pain) to 10 (pain as bad as you can imagine) is recorded on a subject diary twice daily for 5 days before a study visit. The score for each visit is calculated as the mean pain of the 5 diary days morning and evening scores. For each subject, the change in pain will be calculated as the mean pain score at Month 3 minus the mean pain score at Baseline. A negative change value represents a lowering of the pain score (an improvement, or reduction in pain).
Time Frame: 3 Month
Population: 2 of the 3 randomized participants did not complete the follow-up or provide outcome information. As there was only 1 participant that completed the secondary outcome assessment, no statistical analysis will be presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IT Group (SynchroMed/Intrathecal Morphine Sulfate) | Conventional Medical Management
Number analyzed (Participants) | 1 | 0
units on a scale | -3.3 (0) |

3. Secondary Outcome: Opioid-Related Side Effects
Description: Summarize the changes from Baseline to Month 3 between the IT group and CMM group in Common Terminology Criteria for Adverse Events (CTCAE) toxicity score. (from the National Cancer Institute) A subset of 23 specific items of the CTCAE v4.03 were evaluated. The subset was chosen as these criteria were most related to opioid side effects that are of interest in this study. The investigator scored the assessment at each visit. The total score for a visit is based on the sum of 23 individual CTCAE's. The individual scales have a range of 0 to 2, 0 to 3, or 0 to 5 and the total score ranges from 0 (best case) to 90 (worst case). For each subject, the change in toxicity will be calculated as the total toxicity score at Month 3 minus the total toxicity score at Baseline. A negative change value represents a lowering of the subjects toxicity score (an improvement, or reduction in toxicity).
Time Frame: 3 Month
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IT Group (SynchroMed/Intrathecal Morphine Sulfate) | Conventional Medical Management
Number analyzed (Participants) | 1 | 0
units on a scale | -6 (0) |

4. Other Pre Specified Outcome: Sleep Assessment
Description: Compare changes from Baseline to Month 3 between the IT group and CMM group for Apnea-Hypopnea Index (AHI). The AHI was collected via overnight sleep lab polysomnography. The AHI is an index used to indicate the severity of sleep apnea. It is represented by the number of apnea and hypopnea events per hour of sleep. The AHI values for adults are categorized as Normal: AHI<5, Mild sleep apnea: 5≤AHI<15, Moderate sleep apnea: 15≤AHI<30, Severe sleep apnea: AHI≥30. For each subject, the change in AHI will be calculated as the AHI at Month 3 minus the AHI at Baseline. A negative change value represents a lowering of the subjects AHI (an improvement, or reduction in sleep apnea).
Time Frame: 3 Month
Population: 2 of the 3 randomized participants did not complete the follow-up or provide outcome information. As there was only 1 participant that completed the outcome assessment, no statistical analysis will be presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IT Group (SynchroMed/Intrathecal Morphine Sulfate) | Conventional Medical Management
Number analyzed (Participants) | 1 | 0
units on a scale | -10.4 (0) |

ADVERSE EVENTS:
Time Frame: throughout the study duration, from enrollment to 3 months follow-up after implant, an average of 4 months
Arm/Group | IT Group (SynchroMed/Intrathecal Morphine Sulfate) | Conventional Medical Management
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 1/3 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IT Group (SynchroMed/Intrathecal Morphine Sulfate) (N=3) | Conventional Medical Management (N=0)
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0

LIMITATIONS AND CAVEATS:
Due to the small sample size (only 1 IT Group and 0 CMM Group participants completed the primary outcome assessment), statistical tests cannot be performed and conclusions cannot be made on any of the original study objectives.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restrictions on the PI allow for the sponsor to review results communications prior to public release and to embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to sponsor for review. The sponsor is also allowed to require changes for technical correctness and to protect confidential information, copyrightable or patentable material; and when reasonably requested, extend the embargo up to an additional 90 days.